CLINICAL TRIAL: NCT06824467
Title: A Phase 3, Randomized, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Sacituzumab Tirumotecan Maintenance Treatment With or Without Bevacizumab Versus Standard of Care After Second-line Platinum-based Doublet Chemotherapy in Participants With Platinum-sensitive Recurrent Ovarian Cancer (TroFuse-022/ENGOT-ov84/GOG-3103)
Brief Title: A Study to Evaluate the Efficacy and Safety of Sacituzumab Tirumotecan (MK-2870) Treatment Versus Standard of Care in Participants With Platinum-sensitive Recurrent Ovarian Cancer (MK-2870-022/TroFuse-022/ENGOT-ov84/GOG-3103)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-022; MK-2870-022 (Other: MSD); TroFuse-022 (Other: MSD); 2023-508015-23-00 (Registry Identifier: EU CT); U1111-1297-4489 (Registry Identifier: UTN); GOG-3103 (Other: Gynecologic Oncology Group); ENGOT-ov84 (Other: European Network of Gynaecological Oncological Trial Groups (ENGOT)); jRCT2031240722 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab; Histamine Antagonists; Histamine H2 Antagonists; Acetaminophen; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Sacituzumab tirumotecan + Bevacizumab (Experimental): Participants receive 4 mg/kg of sacituzumab tirumotecan once every 2 weeks (Q2W) plus 15 mg/kg of bevacizumab once every 3 weeks (Q3W) via intravenous (IV) infusion over 6 weeks
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Bevacizumab; Drug: H1 receptor antagonist; Drug: H2 receptor antagonist; Drug: Acetaminophen (or equivalent); Drug: Dexamethasone (or equivalent); Drug: Steroid mouthwash (dexamethasone or equivalent)
- Part 2: Sacituzumab tirumotecan (Experimental): Participants receive 4 mg/kg of sacituzumab tirumotecan Q2W via IV infusion until progressive disease or discontinuation. At the physician's discretion, participants receive 15 mg/kg of bevacizumab Q3W via IV infusion until progressive disease or discontinuation.
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Bevacizumab; Drug: H1 receptor antagonist; Drug: H2 receptor antagonist; Drug: Acetaminophen (or equivalent); Drug: Dexamethasone (or equivalent); Drug: Steroid mouthwash (dexamethasone or equivalent)
- Part 2: Standard of care (SOC) (Active Comparator): Participants receive local standard of care until progressive disease or discontinuation. At the physician's discretion, participants receive 15 mg/kg of bevacizumab Q3W via IV infusion until progressive disease or discontinuation.
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — IV Infusion
  Other Names: MK-2870; sac-TMT; SKB264
  Arms: Part 1: Sacituzumab tirumotecan + Bevacizumab; Part 2: Sacituzumab tirumotecan
Biological: Bevacizumab — IV Infusion
  Other Names: Avastin; Altusan; MVASI
Drug: H1 receptor antagonist — Rescue medication taken per approved product label before sacituzumab tirumotecan
  Arms: Part 1: Sacituzumab tirumotecan + Bevacizumab; Part 2: Sacituzumab tirumotecan
Drug: H2 receptor antagonist — Rescue medication taken per approved product label before sacituzumab tirumotecan
  Arms: Part 1: Sacituzumab tirumotecan + Bevacizumab; Part 2: Sacituzumab tirumotecan
Drug: Acetaminophen (or equivalent) — Rescue medication taken per approved product label before sacituzumab tirumotecan
  Arms: Part 1: Sacituzumab tirumotecan + Bevacizumab; Part 2: Sacituzumab tirumotecan
Drug: Dexamethasone (or equivalent) — Rescue medication taken per approved product label before sacituzumab tirumotecan
  Arms: Part 1: Sacituzumab tirumotecan + Bevacizumab; Part 2: Sacituzumab tirumotecan
Drug: Steroid mouthwash (dexamethasone or equivalent) — Rescue medication taken orally 4 times daily
  Arms: Part 1: Sacituzumab tirumotecan + Bevacizumab; Part 2: Sacituzumab tirumotecan

SUMMARY:
The main goals of this study are to learn about the safety of sacituzumab tirumotecan with bevacizumab and if people tolerate it; and If people who take sacituzumab tirumotecan with or without bevacizumab live longer without the cancer getting worse than those who receive standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Has received 4 or more cycles of platinum-based doublet chemotherapy in first-line and a total of 6 cycles of carboplatin-based doublet chemotherapy in second-line setting for ovarian cancer (OC).
* Has platinum-sensitive epithelial OC,
* Has provided tissue of a tumor lesion that was not previously irradiated
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy
* Participants who are hepatitis B surface antigen positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to allocation (Part 1) or randomization (Part 2)
* Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Has an ECOG performance status of 0 to 1 assessed within 7 days before allocation (Part 1) or randomization (Part 2)

Exclusion Criteria:

* Has nonepithelial cancers (germ cell tumors and sex cord-stromal tumors), borderline tumors (low malignant potential), mucinous, seromucinous that is predominantly mucinous, malignant Brenner's tumor and undifferentiated carcinoma
* Has platinum-resistant OC or platinum-refractory OC
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing.
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has received more than 2 prior lines of systemic therapy for OC.
* Has received prior systemic anticancer therapy within 3 weeks or 5 half-lives (whichever is shorter) before allocation (Part 1) or randomization (Part 2)
* Has received prior radiotherapy within 2 weeks of allocation (Part 1) or randomization (Part 2), or has radiation related toxicities, requiring corticosteroids
* Has an additional malignancy that is progressing or has required active treatment within the past 3 years
* Has active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active infection requiring systemic therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2029-04-27 (Estimated); Study Completion 2032-10-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with one or more adverse events (AEs) | Up to 6 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Part 1: Number of participants who discontinue study intervention due to an AE | Up to 6 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Part 2: Progression-free Survival (PFS) | Up to approximately 4 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.

SECONDARY OUTCOMES:
Part 2: Overall Survival (OS) | Up to approximately 4 years
  OS is defined as the time from randomization to death due to any cause
Part 2: Number of participants with one or more AEs | Up to approximately 4 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Part 2: Number of participants who discontinue study intervention due to an AE | Up to approximately 4 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Part 2: Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status-Quality of Life Score | Baseline and up to approximately 4 years
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to Item 30 (""How would you rate your overall quality of life during the past week?") is scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher value indicates a better level of function. The change from baseline in EORTC QLQ-C30 Item 30 score will be reported.
Part 2: Change from Baseline in EORTC QLQ-C30 Physical Functioning Score | Baseline and up to approximately 4 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of physical functioning.
Part 2: Change from Baseline in EORTC QLQ-C30 Role Functioning Score | Baseline and up to approximately 4 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and " Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate a more impaired level of role functioning. Change from baseline in the role functioning score will be presented.
Part 2: Change from Baseline in EORTC Quality of Life Questionnaire-Ovarian Cancer Module 28 (QLQ-OV28) abdominal/gastrointestinal (GI) symptom scale | Baseline and up to approximately 4 years
  The EORTC QLQ-OV28 is an OC-specific, and psychometrically and clinically validated module to supplement the EORTC QLQ-C30. The EORTC QLQ-OV28 abdominal/GI symptom scale is scored on a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (70):
- United States (15):
  - Mount Sinai Cancer Center ( Site 0078), Miami Beach, Florida
  - Sarasota Memorial Hospital ( Site 0075), Sarasota, Florida
  - Florida Cancer Specialists East ( Site 7000), West Palm Beach, Florida
  - St. Dominic's Hospital ( Site 0064), Jackson, Mississippi
  - Nebraska Methodist Hospital ( Site 0053), Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey ( Site 0071), New Brunswick, New Jersey
  - FirstHealth Cancer Center ( Site 0079), Pinehurst, North Carolina
  - University of Cincinnati Medical Center ( Site 0090), Cincinnati, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0056), Tulsa, Oklahoma
  - Oncology Associates of Oregon, P.C.(Willamette Valley Cancer Institute) (WVCI) ( Site 8010), Eugene, Oregon
  - Women & Infants Hospital ( Site 0050), Providence, Rhode Island
  - Texas Oncology - Central/South Texas ( Site 8009), Austin, Texas
  - Texas Oncology - DFW ( Site 8001), Fort Worth, Texas
  - Texas Oncology - San Antonio ( Site 8005), San Antonio, Texas
  - Texas Oncology - Gulf Coast ( Site 8003), Webster, Texas
- Australia (4):
  - Blacktown Hospital ( Site 0211), Sydney, New South Wales
  - Gallipoli Medical Research Ltd ( Site 0214), Brisbane, Queensland
  - Epworth Freemasons ( Site 0217), East Melbourne, Victoria
  - Frankston Hospital ( Site 0216), Frankston, Victoria
- UZ Leuven ( Site 0301), Leuven, Vlaams-Brabant, Belgium
- IBCC - Núcleo de Pesquisa e Ensino ( Site 0424), São Paulo, Brazil
- Colombia (3):
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0806), Bogotá, Bogota D.C.
  - Instituto Nacional De Cancerologia ( Site 0807), Bogotá, Bogota D.C.
  - Oncologos Del Occidente ( Site 0805), Pereira, Risaralda Department
- Denmark (3):
  - Herlev Hospital ( Site 0903), Herlev, Capital Region
  - Aalborg Universitetshospital ( Site 0901), Aalborg, North Denmark
  - Vejle Sygehus ( Site 0902), Vejle, Region Syddanmark
- Finland (2):
  - Kuopion Yliopistollinen Sairaala ( Site 1004), Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala ( Site 1002), Tampere, Pirkanmaa
- France (3):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest ( Site 1101), Bordeaux, Aquitaine
  - Pôle Santé Léonard de Vinci ( Site 1112), Chambray-lès-Tours, Indre-et-Loire
  - Sainte Catherine Institut du Cancer Avignon Provence ( Site 1105), Avignon, Vaucluse
- Israel (2):
  - Rambam Health Care Campus ( Site 1402), Haifa
  - Shaare Zedek Medical Center ( Site 1405), Jerusalem
- Italy (3):
  - Instituto Tumori Giovanni Paolo II ( Site 1505), Bari
  - Istituto Oncologico Veneto IRCCS ( Site 1508), Padua
  - Ospedale Mauriziano ( Site 1509), Torino
- Japan (9):
  - National Hospital Organization Shikoku Cancer Center ( Site 1631), Matsuyama, Ehime
  - Kurume University Hospital ( Site 1640), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 1630), Ōta, Gunma
  - Iwate Medical University Hospital ( Site 1635), Shiwa-gun, Iwate
  - Saitama Medical University International Medical Center ( Site 1632), Hidaka, Saitama
  - Cancer Institute Hospital of JFCR ( Site 1639), Koto, Tokyo
  - Keio University Hospital ( Site 1636), Shinjyuku, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 1628), Fukuoka
  - Niigata Cancer Center Hospital ( Site 1633), Niigata
- IPOR Instituto Peruano de Oncología & Radioterapia ( Site 3604), Lima, Peru
- Romania (2):
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 2215), Cluj-Napoca, Cluj
  - Cabinet Medical Oncomed ( Site 2217), Timișoara, Timiș County
- South Korea (5):
  - National Cancer Center ( Site 2305), Goyang-si, Kyonggi-do
  - Severance Hospital ( Site 2302), Seodaemun-Gu, Seoul
  - Asan Medical Center ( Site 2304), Songpa-gu, Seoul
  - Seoul National University Hospital ( Site 2301), Seoul
  - Samsung Medical Center ( Site 2303), Seoul
- Spain (11):
  - Institut Català d'Oncologia (ICO) - Girona ( Site 2402), Girona, Gerona
  - Hospital General Gregorio Maranon de Madrid ( Site 2412), Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra ( Site 2407), Madrid, Madrid, Comunidad de
  - Hosp Clinico Universitario de Valencia ( Site 2401), Valencia, Valenciana, Comunitat
  - Hospital Vall D Hebron ( Site 2403), Barcelona
  - Hospital Clinic I Provincial de Barcelona ( Site 2409), Barcelona
  - ICO L Hospitalet ( Site 2408), Barcelona
  - Hospital Universitario Reina Sofia ( Site 2406), Córdoba
  - Hospital Ramon y Cajal ( Site 2405), Madrid
  - Hospital Clinico San Carlos... ( Site 2410), Madrid
  - Hospital Universitario 12 de Octubre ( Site 2411), Madrid
- Taiwan (5):
  - Taichung Veterans General Hospital ( Site 2603), Taichung
  - National Cheng Kung University Hospital ( Site 2602), Tainan
  - National Taiwan University Hospital ( Site 2601), Taipei
  - Mackay Memorial Hospital ( Site 2604), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 2605), Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/